CLINICAL TRIAL: NCT07082413
Title: Application of a Frequency Measurement System for Measuring Nutritional Biomarkers: Effects of a Nutritional Intervention on Satisfaction and Improvement in Quality of Life
Brief Title: Biofrequency-Guided Nutrition in Spanish Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Especialidades Espiritu Santo (Other)
Collaborators: Universidad de Almeria (Other); Universidad de Granada (Other); Universidad de Los Lagos (Other); Universidad Loyola Andalucia (Other)
Responsible Party: Principal Investigator, José Francisco López Gil, Investigador principal, Universidad de Especialidades Espiritu Santo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: UALBIO2025/010
Record Dates: First submitted 2025-07-02; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Biofrequency-Guided Nutrition
Keywords: Biofrequency analysis; biomarker-based nutrition; dietary habits; mediterranean diet; nutritional biomarkers; nutritional intervention; young athletes
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard diet (Experimental): The experimental group will undergo a standardized and comprehensive nutritional intervention designed to optimize health outcomes and improve the biomarkers under study. This intervention will incorporate both practical dietary guidelines and an educational component aimed at enhancing participants' understanding of underlying health principles. Participants will receive detailed documentation, including: (1) dietary guidelines outlining the nutritional protocol, (2) a sample monthly meal plan, (3), a structured shopping list, (4) selected recipes and (5) visual meal preparation guides. To facilitate self-monitoring, a food intake log will be provided for daily dietary tracking. The intervention will include an educational program covering key health concepts relevant to the study. Through informational materials and group sessions, participants will receive instruction on topics such as stress physiology, epigenetic mechanisms, chronic disease prevention, and mindful eating pr
  Interventions: Other: Nutritional Intervention
- Usual diet (No Intervention): The control group will maintain their habitual dietary patterns without receiving intervention materials or support. This approach will ensure that all experimental group participants receive identical guidelines, benefiting from multiple modalities of education and support, thereby establishing a robust framework for dietary modification.

INTERVENTIONS:
Other: Nutritional Intervention — This study will follow a randomized controlled trial design aimed at evaluating the impact of nutritional intervention on personal satisfaction and perceived quality of life. The protocol includes two assessment points: a baseline measurement at the start of the intervention (Day 0) and a second measurement after a follow-up period (Day 90), allowing for the analysis of with-in-subject changes associated with the intervention.
  Arms: Standard diet

SUMMARY:
The goal of this clinical trial is to evaluate the feasibility, acceptability, and preliminary efficacy of a biofrequency-guided nutritional intervention in promoting a healthy diet, improving dietary behaviors, and enhancing user satisfaction among healthy Spanish adults. The present study aims to address four main objectives: (1) to analyze the utility of the biofrequency system for non-invasive functional estimates of nutritional status; (2) to evaluate the effectiveness of the associated algorithm in generating bi-omarker-informed dietary recommendations; (3) to assess user and healthcare profes-sional acceptance and satisfaction with the tool; and (4) to examine the effects of the intervention on eating habits.

DETAILED DESCRIPTION:
Background: Biomarker-based nutrition has demonstrated superior efficacy compared to population-level approaches in improving health outcomes. Biofrequency analysis, a non-invasive technique based on the detection of electromagnetic vibrational patterns in hair follicles, offers a promising avenue for rapid functional assessment of nutritional status and epigenetic signals without reliance on blood or urine sampling. Objective: To evaluate the feasibility, acceptability, and preliminary efficacy of a biofrequency-guided nutritional intervention in promoting a healthy diet, improving dietary behaviors, and enhancing user satisfaction among healthy Spanish adults. Methods: In this randomized controlled trial, 154 adults from the Grupo Alcaraz Sport Association (Region of Murcia, Spain) will be allocated to an experimental group receiving individualized lifestyle recommendations based on S-Drive biofrequency analysis and to a control group with no intervention. Participants in the experimental arm will apply tailored dietary guidance over 90 days. Conclusion: This study will generate foundational evidence on the utility of biofrequency technology for precision nutrition. If positive, the findings may inform scalable, low-risk strategies for personalized dietary interventions in preventive and community health settings.

ELIGIBILITY:
Inclusion Criteria:

* No diagnosed chronic illnesses.
* Provision of written informed consent.

Exclusion Criteria:

* Diagnosed chronic illnesses
* No provision of written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-12-07 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Functional Epigenetic Optimization | On day 0 and day 90
  Functional status will be assessed with the S-Drive optimization report, which analyzes resonance frequency patterns from hair follicle samples using proprietary algorithms. The report classifies each participant's physiological functioning into 12 domains grouped into four categories: (1) Micronutrient indicators (vitamins, minerals, amino acids, fatty acids, antioxidants); (2) Systemic physiological indicators (immune system, gut health, circulatory function); (3) Epigenetic and environmental stressors (EMF, ELF radiation, toxins, additives); and (4) Dietary guidance (food choices, hydration, supplementation).
  Each domain is rated on four qualitative levels: "not flagged" (0), "to be considered" (1), "advisable" (2), and "priority" (3). Two derived scores will be analyzed: the total number of "priority" domains and a cumulative optimization score (0-36). These will be used to assess within-subject changes and between-group differences from baseline to follow-up.

SECONDARY OUTCOMES:
Anthropometric Data | On day 0 and day 90
  Anthropometric data, including current body weight (in kilograms) and height (in centimeters), will be self-reported by participants. These measurements will be used to compute body mass index (BMI), which is calculated by dividing weight in kilograms by the square of height in meters (kg/m²). BMI categories will be defined in accordance with World Health Organization (WHO) standards: BMI < 18.5 ("underweight"), 18.5 ≤ BMI < 24.9 ("normal weight"), 25 ≤ BMI < 29.9 ("overweight"), 30 ≤ BMI < 34.9 ("obesity class I"), 35 ≤ BMI < 39.9 ("obesity class II"), and BMI ≥ 40 ("obesity class III") (Weir & Jan, 2023). Although self-reported measurements may be susceptible to bias, previous research indicates that self-reported BMI estimates are generally valid in adult populations (Stommel & Schoenborn, 2009).
24-Hour Movement Behaviors | On day 0 and day 90
  Physical activity across work/school, transport, and leisure will be assessed with the validated PAS-2.1S (Valles-Medina et al., 2021). The scale has nine items: six on daily activities (weekday/weekend sleep, sedentary behavior, active physical activity, leisure, commuting) and three on weekly activities. Sleep duration is self-reported; sedentary behavior covers commuting by car/public transport and screen/reading time. The weekly subscale records light (e.g., walking), moderate (e.g., gardening), and vigorous (e.g., running) activities. Activity intensity, based on METs (Ainsworth et al., 2000), includes values such as sleep (0.9), sitting work (1.5), light activity (3.0), and vigorous activity (6.0). Daily work/transport METs are multiplied by five; sleep/leisure by seven. Missing daily hours (<24) are doubled. Total METs from daily and weekly activities yield total energy expenditure.
Adherence to the Mediterranean diet (MedDiet) | On day 0 and day 90
  Adherence to the Mediterranean diet (MedDiet) will be measured using the PREvención con DIeta MEDiterránea (PREDIMED) questionnaire (Martínez-González et al., 2012). Participants will report the frequency or quantity of consumption of 12 core dietary components (e.g., fruits, vegetables, olive oil, nuts) and two related dietary habits. The 14-item tool assigns binary scores (0 or 1) to each component, with total scores ≥9 indicative of high adherence to the MedDiet.
Tobacco smoking | On day 0 and day 90
  Tobacco use will be assessed with two questions. First, participants will be asked: "Have you ever smoked tobacco in your lifetime?", with response options ranging from (a) never to (g) 30 times or more. Second, adolescents will be asked about current smoking frequency: (a) I do not smoke, (b) less than once a week, (c) more than once a week but not daily, and (d) every day.
Alcohol consumption | On day 0 and day 90
  Alcohol consumption will be assessed with: "Have you ever consumed alcohol in your lifetime?", offering options: never, once or twice, 3-5, 6-9, 10-19, 20-29, and 30+ times. Additionally, participants will report the frequency of different alcoholic beverages, coded into days per week: never (0), almost never (0.10), monthly (0.25), weekly (1), daily (7). The mean weekly frequency will then be calculated. Based on these data, participants will be classified as non-drinkers (never consumed alcohol), regular drinkers (weekly or more), or irregular drinkers (monthly or less). Binge drinking will be measured by asking: "Have you ever consumed enough alcohol to become intoxicated?", with options: never, once, 2-3, 4-10, and more than 10 times. Excessive consumption will be defined as having become intoxicated on at least one occasion.
Cannabis use | On day 0 and day 90
  Cannabis consumption will be assessed with the question: "Have you ever used cannabis in your lifetime?", using response options: (a) never, (b) once or twice, (c) 3 to 5 times, (d) 6 to 9 times, (e) 10 to 19 times, (f) 20 to 29 times, and (g) 30 times or more.
Depressive Symptoms | On day 0 and day 90
  Depressive symptoms will be measured using the Spanish version of the Beck Depression Inventory-II (BDI-II) (Sanz & Navarro, 2003). This self-administered instrument consists of 21 items, each with four response options representing increasing severity over the preceding two weeks. Item scores range from 0 to 3, yielding a total score between 0 and 63.
Anxiety Symptoms | On day 0 and day 90
  Anxiety symptoms will be evaluated using the Generalized Anxiety Disorder-7 (GAD-7) questionnaire, validated for primary care (Löwe et al., 2008). This instrument contains seven items (Spitzer et al., 2006), assessing symptoms such as nervousness, worry, restlessness, and irritability over the previous 14 days. Items are rated on a four-point Likert scale: never (0 points), several days (1 point), half of the days (2 points), and almost every day (3 points). Total scores range from 0 to 21, with thresholds as follows: no anxiety (0-4 points), mild anxiety symptoms (5-9 points), moderate anxiety symptoms (10-14 points), and severe anxiety symptoms (15-21 points).
Perceived stress | On day 0 and day 90
  Perceived stress will be assessed using the Spanish version of the Perceived Stress Scale-14 (PSS-14) (Remor, 2006; Remor & Carrobles, 2001). This 14-item instrument utilizes a five-point response scale: never (0 points), almost never (1 point), once in a while (2 points), often (3 points), and very often (4 points). The total score is calculated by reversing the responses for items 4, 5, 6, 7, 9, 10, and 13 using the conversion scale (0=4, 1=3, 2=2, 3=1, 4=0) and then summing the scores of all 14 items. Higher scores reflect greater perceived stress.
Disordered eating | On day 0 and day 90
  Disordered eating behaviors will be evaluated using the Sick, Control, One, Fat, Food (SCOFF) questionnaire, a concise and validated screening instrument designed to identify individuals at risk for eating disorders (Garcia-Campayo et al., 2005). The SCOFF consists of five items that capture core dimensions of disordered eating, including restrictive intake, preoccupation with weight and shape, and compensatory behaviors. Each item requires a binary (yes/no) response, and a score of ≥2 affirmative answers indicate an increased risk for an eating disorder.

OTHER OUTCOMES:
Sociodemographic Data | On day 0
  Participants will provide self-reported information regarding their sex and age. Data will also be gathered on their current engagement in educational pursuits, employment status, participation in remunerated activities, and their specific occupation. Additionally, participants will be asked to indicate the primary reason for their most recent visit to primary care services. Educational attainment will be categorized as follows: (a) incomplete primary education (<6 years), (b) completed primary education (6 years), (c) incomplete secondary education (<4 years), (d) completed secondary education (4 years), (e) incomplete higher education (<2 years of baccalaureate studies), and (f) completed higher education (2 years of baccalaureate studies or a bachelor's degree).

IPD SHARING:
Plan to Share IPD: No
IPD (Individual Participant Data) will not be shared because the study involves sensitive human data protected under the General Data Protection Regulation (GDPR). Additionally, the biological data are generated through a proprietary device and algorithm (S-Drive, Cell Wellbeing) that are subject to confidentiality agreements, which prevent the release of raw data. As this is an exploratory randomized controlled trial, there is also no current plan for public data sharing.